CLINICAL TRIAL: NCT07297758
Title: Investigation of Latissimus Dorsi Muscle Activation During Shoulder Extension Exercises
Brief Title: Latissimus Dorsi Activation During Shoulder Extension Exercises
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, Professor, Department of Physiotherapy and Rehabilitation, Hacettepe University
Other Study IDs: Shoulder-EX-EMG
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Muscle Activation
Keywords: Shoulder; Latissimus Dorsi; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Active Adults: Ages 18-40; Tegner ≥5; no GH restriction; no shoulder/cervical/lumbar complaints in last 6 months; no systemic/neurologic disease; BMI ≤25 kg/m².
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Standing with the shoulder in ~30° abduction and external rotation and the elbow extended, participants elevate the arm to three preset flexion angles (30°,60°, 90°, 120°; measured by goniometer) and then perform shoulder extension past the trunk against color-coded elastic bands. Bands are anchored overhead and pulled diagonally downward; the band angle is adjusted to match each shoulder-flexion condition. Tempo is metronome-paced: 3 s concentric, 3 s isometric (at peak), 3 s eccentric. Resistance is individualized using the OMNI Perceived Exertion Scale and titrated until 6-8/10 is reached prior to data capture. Each condition is recorded for 3 repetitions with ~5 s between reps; ~2 min rest is provided between conditions. A brief familiarization (~3 min per condition) is given, and the order of MVICs and exercise conditions is randomized.

SUMMARY:
This observational, cross-sectional laboratory study at Hacettepe University will examine surface EMG activation of the latissimus dorsi during resisted, dynamic shoulder extension performed at three shoulder flexion angles (30°,60°, 90°, 120°). The primary objective is to quantify latissimus dorsi activation and to determine how elevation angle influences activation; secondary analyses compare synergists.

DETAILED DESCRIPTION:
During shoulder abduction or flexion, narrowing of the subacromial space can lead to subacromial pain syndrome. Weakness or poor coordination of the scapulothoracic and scapulohumeral muscles is among the main causes of subacromial narrowing in individuals with symptomatic rotator cuff tendinopathy. More specifically, insufficient scapular upward rotation and posterior tilt, together with an inadequate ability of the rotator cuff to counter the deltoid's superior pull on the humeral head, may cause impingement of the subacromial soft tissues during overhead dynamic tasks. In young, healthy shoulders, the cranially directed forces that occur during abduction are balanced by co-contraction of the rotator cuff, which prevents superior translation of the humeral head and protects subacromial tissues. When this stabilizing role of the rotator cuff diminishes, the deltoid attempts to compensate; however, this compensation produces a more cranially oriented force, increasing superior migration of the humeral head and the likelihood of subacromial pain.

The latissimus dorsi (LD) originates from the spinous processes of the lower thoracic vertebrae, the thoracolumbar fascia, and the iliac crest, and-together with the teres major-attaches to the medial lip of the intertubercular groove of the humerus. It contributes to shoulder adduction, internal rotation, and extension, and is an important muscle directly linking the upper limb to the trunk. In addition to the rotator cuff, the glenohumeral adductors (pectoralis major and latissimus dorsi) also help limit superior translation of the humeral head; owing to the medio-inferior direction of their tendon force vectors, they act as humeral head depressors. Osteokinematically, the LD can pull the humeral head inferiorly over the glenoid fossa, potentially helping to prevent subacromial impingement.

Various exercises have been recommended for LD rehabilitation, and surface electromyography (sEMG) studies have examined LD activity during movements such as pulldown and pullover. Numerous studies have also sought to determine maximal voluntary isometric contraction (MVIC) of the LD. Prior EMG research indicates that the highest LD MVIC levels are obtained during maximal isometric shoulder extension. A recent study using both surface and fine-wire electrodes also recorded higher LD activation during shoulder extension compared with trunk tasks. Although shoulder extension exercises are widely used at different elevation angles in clinical practice, the effects of performing extension at different angles-particularly on LD activation-have not been clearly delineated. Despite various recommendations for LD rehabilitation, it remains unclear whether different implementations produce different activation profiles, and LD activation during dynamic application of this exercise has not yet been investigated. Therefore, it is important to examine how the highest LD activity obtained during maximal isometric shoulder extension changes when the exercise is performed dynamically. Defining the LD activation profile in dynamic exercise may inform appropriate exercise selection in clinical rehabilitation and help reduce the risk of subacromial impingement.

Aim. To address this gap by examining the level of LD activation during dynamic shoulder extension relative to the reference activity determined by maximal isometric shoulder extension. The study has two specific aims: (1) to determine the EMG activation level of the latissimus dorsi during a shoulder extension exercise, and (2) to investigate the effects of performing shoulder extension at different elevation angles on latissimus dorsi activation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40,
* No restriction of the glenohumeral joint,
* No complaints related to the shoulder, cervical, or lumbar region in the last 6 months,
* No systemic or neurological disease,
* Agreeing to participate in the study,
* A Tegner Activity Score of 5 or higher,

Exclusion Criteria:

* A body mass index greater than 25 kg/m2

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, physically active adults aged 18-40 years, recruited from a university cohort and local community, for a single-visit laboratory EMG study at Hacettepe University. Eligibility requires Tegner ≥5, full glenohumeral range of motion, no shoulder/cervical/lumbar complaints in the past 6 months, and no systemic or neurological disease; individuals with BMI >25 kg/m² are excluded
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Electromyography | Baseline (Day 1)
  Muscle activation will be assessed with an 8-channel surface EMG system (TeleMyo DTS, Noraxon). Following SENIAM, bipolar Ag/AgCl electrodes (2 cm inter-electrode distance) will be placed over medial and lateral latissimus dorsi, teres major, infraspinatus, posterior deltoid, and triceps brachii, secured with double-sided tape. Before exercise, MVICs will be obtained on the dominant arm by the same assessor (3 × 5 s with 30 s between trials and 2 min between muscles) using standardized, literature-based positions with verbal encouragement.The exercise protocol will consist of elastic-band resisted shoulder extension performed for three repetitions (3 s concentric-3 s isometric-3 s eccentric) with 5 s between repetitions and 2 min rest between conditions, while EMG from all target muscles is recorded and timing is controlled by a metronome.

SECONDARY OUTCOMES:
Activity Level | Baseline (Day 1)
  Baseline physical activity will be characterized using the Tegner Activity Scale (0-10) prior to testing; higher scores indicate greater habitual activity.

CONTACTS AND LOCATIONS:
Overall Officials: Irem Duzgun, PhD, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samandag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. De-identified aggregate results will be disseminated in publications. The dataset includes physiological signals; synchronized videos are deleted after analysis.